CLINICAL TRIAL: NCT02331108
Title: A Comparison of the Effect on Temperature Between Patients Induced With Intravenous Propofol vs Inhalation Induction With Sevoflurane
Brief Title: A Comparison of Inhalation vs. Intravenous Induction
Acronym: INHvsIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Jonathan Roth, Staff Anesthesiologist, M.D., Albert Einstein Healthcare Network
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HN4613
Record Dates: First submitted 2014-11-20; First posted 2015-01-06 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia | interventions — Anesthesia; Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- sevoflurane in 100% oxygen, age <56 (Active Comparator): The intervention will be the randomized selection of anesthetic induction technique to sevoflurane in 100% oxygen and temperatures will be recorded per protocol. Age 18-55.
  Interventions: Drug: Selection of anesthetic induction technique
- sevoflurane in 50% nitrous, age <56 (Active Comparator): The intervention will be the randomized selection of anesthetic induction technique to sevoflurane in 50% oxygen and 50% nitrous oxide. Age 18-55.
  Interventions: Drug: Selection of anesthetic induction technique
- propofol, age <56 (Active Comparator): The intervention will be the randomized selection of anesthetic induction technique to intravenous induction with 2.2 mg/kg propofol. Age 18-55.
  Interventions: Drug: Selection of anesthetic induction technique
- propofol with phenylephrine, age <56 (Active Comparator): The intervention will be the randomized selection of anesthetic induction technique to intravenous induction 2.2 mg/kg propofol immediately preceded by 160 mcg intravenous phenylephrine. Age 18-55.
  Interventions: Drug: Selection of anesthetic induction technique
- sevoflurane in 100% oxygen, age >55 (Active Comparator): The intervention will be the randomized selection of anesthetic induction technique to sevoflurane in 100% oxygen and temperatures will be recorded per protocol. Age >55.
  Interventions: Drug: Selection of anesthetic induction technique
- sevoflurane in 50% nitrous, age >55 (Active Comparator): The intervention will be the randomized selection of anesthetic induction technique to sevoflurane in 50% oxygen and 50% nitrous oxide. Age >55.
  Interventions: Drug: Selection of anesthetic induction technique

INTERVENTIONS:
Drug: Selection of anesthetic induction technique — Standard anesthesia care will be provided after induction based on randomization. Temperatures will be monitored every 15 minutes
  Other Names: anesthesia, anesthetic induction, sevoflurane, propofol

SUMMARY:
To compart differences on the effect on core temperature between anesthetic induction with intravenous propofol versus inhalation induction with sevoflurane

DETAILED DESCRIPTION:
Hypothermia occurs with anesthetic induction due to redistribution hypothermia. Hypothermia has adverse effects and should be avoided or minimized. Intravenous propofol induction is the most common technique used for anesthetic induction. There is preliminary evidence that there is less redistribution hypothermia when anesthetic induction is achieved by inhalation induction compared to intravenous induction. There is not enough data to compel a change in practice patterns. This study will enroll a larger number of patients in order to provide stronger evidence that there is a significant difference between induction techniques on body temperature. Patients will be randomly assigned to two variation of inhalation induction techniques and two variations of intravenous induction. The effect on temperature between the four groups will be compared. Reducing the degree of hypothermia has the potential to decrease surgical infection rate as well as providing other benefits to patients.

ELIGIBILITY:
Inclusion Criteria:

Elective surgery Adult, age >= 18 years old Scheduled for general anesthesia Medically fit and able to safely go any of the four anesthetic inductions in the study

Exclusion Criteria:

Emergency surgery, or any other aspiration risk Minor, age <18 Pregnant Febrile illness Contraindication to nasal instrumentation Allergy to propofol Malignant hyperthermia Requiring Total Invravenous Anesthesia (TIVA) Inability to oxygenate on less than 50% FiO2 Intra-cranial surgery Receiving vasoactive medications Significant valvular heart disease Unstable cardiac disease Surgery requiring prone or lateral positioning Contraindication to nitrous oxide Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan V Roth, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert EinsteinMedical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Roth JV, Braitman LE, Hunt LH. Induction techniques that reduce redistribution hypothermia: a prospective, randomized, controlled, single blind effectiveness study. BMC Anesthesiol. 2019 Nov 6;19(1):203. doi: 10.1186/s12871-019-0866-8. PMID 31694576

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sevoflurane in 100% Oxygen, Age <56 | Sevoflurane in 50% Nitrous, Age <56 | Propofol, Age <56 | Propofol With Phenylephrine, Age <56 | Sevoflurane in 100% Oxygen, Age >55 | Sevoflurane in 50% Nitrous, Age >55
Started | 51 | 52 | 51 | 51 | 52 | 52
Completed | 50 | 50 | 50 | 50 | 50 | 50
Not Completed | 1 | 2 | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane in 100% Oxygen, Age <56 | Sevoflurane in 50% Nitrous, Age <56 | Propofol, Age <56 | Propofol With Phenylephrine, Age <56 | Sevoflurane in 100% Oxygen, Age >55 | Sevoflurane in 50% Nitrous, Age >55 | Total
Number analyzed (Participants) | 51 | 52 | 51 | 51 | 52 | 52 | 309
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 52 | 51 | 51 | 21 | 25 | 251
  >=65 years | 0 | 0 | 0 | 0 | 31 | 27 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (10.1) | 43.0 (8.8) | 39.0 (11.2) | 40.6 (9.1) | 68.2 (8.4) | 66.2 (7.4) | 50.0 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 20 | 30 | 29 | 19 | 25 | 153
  Male | 21 | 32 | 21 | 22 | 33 | 27 | 156
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51 | 52 | 51 | 51 | 52 | 52 | 309

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Core Temperature
Description: Core temperature at 15 minute intervals
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: degree C
Arm/Group | Sevoflurane in 100% Oxygen, Age <56 | Sevoflurane in 50% Nitrous, Age <56 | Propofol, Age <56 | Propofol With Phenylephrine, Age <56 | Sevoflurane in 100% Oxygen, Age >55 | Sevoflurane in 50% Nitrous, Age >55
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50
degree C
  15 minute temperature | 36.42 (.49) | 36.44 (.44) | 35.96 (.40) | 36.35 (.38) | 36.34 (.46) | 36.41 (.52)
  30 minute temperature | 36.41 (.49) | 36.48 (.44) | 35.95 (.41) | 36.36 (.40) | 36.31 (.48) | 36.38 (.53)
  45 minute temperature | 36.47 (.53) | 36.50 (.43) | 36.00 (.45) | 36.45 (.40) | 36.29 (.50) | 36.41 (.57)
  60 minute temperature | 36.52 (.56) | 36.57 (.42) | 36.03 (.53) | 36.51 (.43) | 36.34 (.51) | 36.44 (.55)

2. Primary Outcome: Temperature Below 36.0 Degrees C
Description: Percentage of patients who had at least one temperature below 36.0 degrees C in the first hour of anesthesia
Time Frame: Intraoperative
Population: Percentage of patients who had one core temperature reading below 36.0 degree C in the first hour of anesthesia
Measure: Number; unit: Percentage
Arm/Group | Sevoflurane in 100% Oxygen, Age <56 | Sevoflurane in 50% Nitrous, Age <56 | Propofol, Age <56 | Propofol With Phenylephrine, Age <56 | Sevoflurane in 100% Oxygen, Age >55 | Sevoflurane in 50% Nitrous, Age >55
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50
Percentage | 8 | 8 | 30 | 8 | 14 | 14

3. Secondary Outcome: Measurement of Blood Pressure
Description: Blood pressure decrease after intravenous anesthetic induction
Time Frame: intraoperative
Population: Percentage of patients whose blood pressure decreased after propofol administration
Measure: Number; unit: percentage of patients
Arm/Group | Propofol, Age <56 | Propofol With Phenylephrine, Age <56
Number analyzed (Participants) | 50 | 50
percentage of patients | 49 | 29

ADVERSE EVENTS:
Arm/Group | Sevoflurane in 100% Oxygen, Age <56 | Sevoflurane in 50% Nitrous, Age <56 | Propofol, Age <56 | Propofol With Phenylephrine, Age <56 | Sevoflurane in 100% Oxygen, Age >55 | Sevoflurane in 50% Nitrous, Age >55
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/51 | 0/51 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/51 | 0/51 | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No